CLINICAL TRIAL: NCT03800784
Title: Study of 18F-DCFPyL PET/CT, for Detection of Radiological Progression in Patients With Metastatic (M+) and Non-metastatic (M0) Castration Resistant Prostate Cancer Receiving Standard Androgen Receptor Targeted Treatment
Brief Title: Study of 18F-DCFPyL PET/CT Imaging in Patients With Prostate Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1863; IRB00150136 (Other: JHM IRB)
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: 18F-DCFPyL PET/CT PyL; PSMA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL Injection (Experimental): A single dose of 9±1 mCi (333±37 MBq) IV injection of 18F-DCFPyL
  Interventions: Drug: 18F-DCFPyL Injection

INTERVENTIONS:
Drug: 18F-DCFPyL Injection — A single dose of 9±1 mCi (333±37 MBq) IV injection of 18F-DCFPyL
  Other Names: PyL

SUMMARY:
This study evaluates the rate of radiological disease progression with the new 2nd generation positron emission tomography (PET) radiopharmaceutical, 18F-DCFPyL, in patients with metastatic castration (mCRPC) and non-metastatic (nmCRPC) castration resistant prostate cancer who have evidence of biochemical (PSA) disease progression without evidence of radiological disease progression on conventional standard radiologic testing (99mTc-methylene diphosphonate bone scan and CT).

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of prostate cancer
* Patients receiving androgen deprivation treatment (ADT) with GnRH analogs, GnRH antagonists or bilateral orchiectomy of any duration.
* Cohort A: nmCRPC (status post- primary treatment with radical prostatectomy, radiation of any type or both)

  * Negative 99mTc-methylene diphosphonate bone scan and CT of the chest abdomen and pelvis within 6 weeks of 18F-DCFPyL PET/CT
  * Treatment with ADT with or without a second line novel AR targeted treatment (abiraterone, enzalutamide, or both) or 4 weeks after discontinuation of first generation antiandrogen (bicalutamide , flutamide, nilutamide- one or more permitted) for ≥ 12 months.
  * Rising PSA ≥ 10 ng/ml (confirmed by 2 determinations one week apart)
  * PSADT ≤ 9 months
* Cohort B: mCRPC

  * Treatment with ADT with or without abiraterone and or enzalutamide or both for ≥ 6 months and/or 4 weeks after discontinuation of first generation antiandrogen (bicalutamide , flutamide, nilutamide- one or more permitted).
  * PSA ≥ 2.0 ng/ml confirmed X 1 week apart, any PSADT
* Patients enrolled in other clinical trials are eligible if they satisfy all other criteria of eligibility.
* No new therapeutic interventions planned or scheduled to be instituted prior to the course of this study both on cohorts A and B before conventional radiologic progression is evidenced.
* Patients or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures.

Exclusion Criteria:

* Patient will be excluded from enrollment if he had a radioisotope within 5 physical half-lives prior to PET imaging

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity 18F-DCFPyL PET/CT imaging to detect metastatic prostate cancer | 3 years
  Proportion of patients demonstrating disease progression by conventional criteria evaluated by CT scan and 99mTc-methylene diphosphonate bone scan and on 18F-DCFPyL PET/CT.

SECONDARY OUTCOMES:
Correlation of findings on 18F-DCFPyL PET/CT with conventional imaging as determined by Number of Lesions detected on each imaging modality | 3 years
  Number of lesions detected on 18F-DCFPyL PET/CT in comparison to number of lesions detected on conventional imaging (99mTc-methylene diphosphonate bone scan and CT)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Markowski, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No